CLINICAL TRIAL: NCT01740024
Title: An Open-label, Multicentre Study Comparing the Biological Potency of the Native, Depigmented and Depigmented Polymerized Cat Epithelial Allergenic Extracts.
Brief Title: Biological Potency of the Cat Epithelial Allergenic Extracts
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Laboratorios Leti, S.L. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 206-PG-PRI-190; 2012-001931-30 (EudraCT Number)
Record Dates: First submitted 2012-11-13; First posted 2012-12-04 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2012-11

CONDITIONS: Cat Allergy (Disorder)
Keywords: Immunotherapy; Subcutaneous immunotherapy; Skin Prick Test; Dose Response Prick Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Dose-Response Skin Prick Tests) (Experimental): 3 different cat epithelium allergenic extracts at 3 different concentrations Positive control Negative control
  Interventions: Biological: 1 (Dose Response Skin Prick Tests)

INTERVENTIONS:
Biological: 1 (Dose Response Skin Prick Tests) — 3 different cat epithelium allergenic extracts at 3 different concentrations, together with a positive and negative control will be tested in every patient in duplicate on the volar surface of the forearm.

SUMMARY:
The primary objective of this clinical trial is to quantify the loss of in vivo biological potency of a depigmented polymerized (DPP) allergenic cat epithelial extract versus the native allergenic extract (N).

DETAILED DESCRIPTION:
This is an open-label, non-randomized phase II clinical trial.

Three different concentrations of three different cat epithelial allergenic extracts, together with a positive and negative control, using 10 mg/ml histamine dihydrochloride and a glycerated phenol saline solution, respectively, will be tested in every subject on the volar surface of the forearm.

ELIGIBILITY:
Inclusion Criteria:

A subject will be eligible for inclusion in the study only if all of the following criteria are met:

* The subject (and/or legal representative, where applicable) has given written, signed and dated informed consent.
* Subjects of either sex and of any race or ethnic group.
* Age > 18 years and < 60 years on the day of inclusion in the study.
* Positive clinical history of allergy to cat epithelia (i.e., rhinitis, conjunctivitis, rhinoconjunctivitis, asthma, urticaria, etc. ).
* A positive prick-test (mean diameter of papule ≥ 3 mm or area of papule ≥ 7 mm2) with a commercial extract of cat epithelium. The results of the prick-test will be valid if they were obtained in the year prior to inclusion of the subject in the study.
* A positive specific IgE test (> 0.70 KU/l) for cat epithelium. The results of the IgE test will be valid if they were obtained in the year prior to inclusion of the subject in the study.

Exclusion Criteria:

A subject will NOT be eligible for inclusion in the study if any of the following criteria are met:

* Immunotherapy in the last 5 years involving allergens known to be able to interfere with the test allergen (e.g., cat extract).
* Use of drugs that can interfere with the skin response before and during the study (e.g., antihistamines), within the intervals established in section 9.1 and appendix 1.
* Treatment with any of the following medicines: tricyclic or tetracyclic antidepressants or MAOIs (Monoamine oxidase inhibitors), beta-blockers or chronic use of oral corticosteroids or use of corticosteroids via either the oral or the parenteral route in repeated and intermittent dosing regimens (> 10 mg/day of prednisone or equivalent).
* Pregnant or nursing women and women with a positive pregnancy test in visit 2.
* Dermographism affecting the skin of the test site, in either of the two visits to the study centre.
* Atopic dermatitis affecting the skin of the test site, in either of the two visits to the study centre.
* Urticaria affecting the skin of the test site, in either of the two visits to the study centre.
* Clinically relevant immune system diseases (both autoimmune disorders and immune deficiencies). (Hashimoto's thyroiditis with hypothyroidism well controlled through thyroid hormone therapy does not necessarily represent a contraindication. Graves' disease (hyperthyroidism) would be an exclusion criterion due to the potential risk in the event adrenaline must be used.)
* Serious uncontrolled diseases that may increase the safety risk of the subjects participating in the study, including but not limited to the following: heart failure, serious or uncontrolled respiratory diseases, endocrine disorders, clinically relevant liver or kidney diseases, or haematological disorders.
* Patents with diseases or conditions that limit adrenaline use (coronary disease, severe arterial hypertension, etc.).
* Serious psychiatric, psychological or neurological problems.
* Medication, alcohol or illegal drug abuse in the last year.
* Participation in any other clinical trial during the 30 days (or 5 times the biological half-life of the investigational product - whichever is longest) prior to inclusion of the subject in this study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2012-11; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Wheal size area (mm2)elicited on the skin after the dose-response prick-test | Test sites should be inspected and recorded 15-20 min after application
  Wheal size area (mm2)elicited on the skin after the dose-response prick-test, in duplicate, of the native and depigmented polymerized cat epithelial allergenic extracts, together with the area of the wheals induced by the positive and negative controls.

SECONDARY OUTCOMES:
Wheal size area (mm2)elicited on the skin after the dose-response prick-test | Test sites should be inspected and recorded 15-20 min after application
  Wheal size area (mm2)elicited on the skin after the dose-response prick-test, in duplicate, of the native and depigmented cat epithelial allergenic extracts, together with the area of the wheals induced by the positive and negative controls.
Wheal siza area (mm2)elicited on the skin after the dose-response prick-test | Test sites should be inspected and recorded 15-20 min after application
  Wheal siza area (mm2)elicited on the skin after the dose-response prick-test, in duplicate, of the depigmented and depigmented polymerized cat epithelial allergenic extracts, together with the area of the wheals induced by the positive and negative controls.
Determine the HEP dose of the native (N) cat epithelial allergenic extract | Wheals will be elicited in visit 2. CRFs will be retrieved, measured in-house and filed back in the site before study closure (maximum 3 months after being elicited).
  Calculation will be made of the 10 HEP dose of the native (N) cat epithelial allergenic extract.
Loss of in vitro potency of the cat epithelial allergenic extracts | Blood will be collected in visit 2. Serum samples will be analyze once every sample is received. The samples will be analyzed at most 12 months after received
  To quantify the loss of in vitro potency of cat epithelial allergenic extracts, based on specific IgE and IgG inhibition studies.

CONTACTS AND LOCATIONS:
Overall Officials: Lena M Erbiti, Study Chair — Laboratorios LETI, S.L.Unipersonal
Locations (2):
- Spain (2):
  - Fundación Jimenez Diaz, Madrid, Madrid / Madrid
  - Hospital El Tomillar - Area Hospitalaria de Valme, Dos Hermanas, Sevilla, Sevilla / Andalucia